CLINICAL TRIAL: NCT02511106
Title: A Phase III, Double-blind, Randomized, Placebo-controlled Multi-centre, Study to Assess the Efficacy and Safety of AZD9291 Versus Placebo, in Patients With Epidermal Growth Factor Receptor Mutation Positive Stage IB-IIIA Non-small Cell Lung Carcinoma, Following Complete Tumour Resection With or Without Adjuvant Chemotherapy (ADAURA).
Brief Title: AZD9291 Versus Placebo in Patients With Stage IB-IIIA Non-small Cell Lung Carcinoma, Following Complete Tumour Resection With or Without Adjuvant Chemotherapy.
Acronym: ADAURA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5164C00001; 2023-506524-82-00 (Registry Identifier: CTIS); 2015-000662-65 (EudraCT Number)
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Stage IB-IIIA Non-small Cell Lung Carcinoma
Keywords: Stage IB-IIA-IIIA Non-Small Cell Lung Cancer; EGFRm+; Ex19Del; L858R; AZD9291; Phase III, adjuvant chemotherapy; complete tumour resection; EGFR-TKI
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD9291 (Experimental): AZD9291 (80 mg or 40 mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: AZD9291 80 mg/40 mg; Drug: Open-label AZD9291 80 mg/40 mg
- Placebo AZD9291 (Placebo Comparator): Matching placebo for AZD9291 (80 mg or 40 mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: Placebo AZD9291 80 mg/40 mg

INTERVENTIONS:
Drug: AZD9291 80 mg/40 mg — The initial dose of AZD9291 80 mg once daily can be reduced to 40 mg once daily.
  Arms: AZD9291
Drug: Placebo AZD9291 80 mg/40 mg — The initial dose of Placebo AZD9291 80 mg once daily can be reduced to 40 mg once daily.
  Arms: Placebo AZD9291
Drug: Open-label AZD9291 80 mg/40 mg — Eligible patients will be offered open-label osimertinib upon recurrence and in the absence of intervening systemic anti-cancer therapy.
  Arms: AZD9291

SUMMARY:
To assess the efficacy and safety of AZD9291 versus Placebo, in patients with Epidermal Growth Factor Receptor Mutation Positive stage IB-IIIA non-small cell lung carcinoma, following complete tumour resection with or without adjuvant chemotherapy

DETAILED DESCRIPTION:
This is a phase 3 double-blind, randomized, placebo-controlled, study to assess the efficacy and safety of AZD9291 versus placebo in patients with stage IB-IIIA non-small cell lung cancer (NSCLC) with centrally confirmed, most common sensitising EGFR mutations (Ex19Del and L858R) either alone or in combination with other EGFR mutations as confirmed by a central test, who have had complete tumour resection, with or without postoperative adjuvant chemotherapy. Adjuvant chemotherapy should have consisted of a platinum based doublet given for a maximum of 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at least 18 years.
2. Histologically confirmed diagnosis of primary non small lung cancer (NSCLC) on predominantly non-squamous histology
3. MRI or CT scan of the brain must be done prior to surgery as it is considered standard of care.
4. Patients must be classified post-operatively as Stage IB, II or IIIA on the basis of pathologic criteria.
5. Confirmation by the central laboratory that the tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations including T790M.
6. Complete surgical resection of the primary NSCLC is mandatory. All gross disease must have been removed at the end of surgery. All surgical margins of resection must be negative for tumour.
7. Complete recovery from surgery and standard post-operative therapy (if applicable) at the time of randomization.
8. World Health Organization Performance Status of 0 to 1.
9. Female patients should be using adequate contraceptive measures, should not be breast feeding, and must have a negative pregnancy test prior to first dose of study drug; or female patients must have an evidence of non-child-bearing potential.

Exclusion Criteria:

1. Treatment with any of the following:

   * Pre-operative or post-operative or planned radiation therapy for the current lung cancer
   * Pre-operative (neo-adjuvant) platinum based or other chemotherapy
   * Any prior anticancer therapy
   * Prior treatment with neoadjuvant or adjuvant EGFR-TKI at any time
   * Major surgery (including primary tumour surgery, excluding placement of vascular access) within 4 weeks of the first dose of study drug
   * Patients currently receiving medications or herbal supplements known to be potent inducers of cytochrome P450 (CYP) 3A4
   * Treatment with an investigational drug within five half-lives of the compound or any of its related material.
2. Patients who have had only segmentectomies or wedge resections
3. History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, or other solid tumours curatively treated with no evidence of disease for > 5 years following the end of treatment.
4. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
5. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
6. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of AZD9291.
7. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 ECGs, using the screening clinic ECG machine-derived QTc value.
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
8. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
9. Inadequate bone marrow reserve or organ function.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2029-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (193):
- United States (23):
  - Research Site, Los Angeles, California
  - Research Site, Santa Monica, California
  - Research Site, Santa Rosa, California
  - Research Site, Torrance, California
  - Research Site, Grand Junction, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Norwalk, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Athens, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Bethesda, Maryland
  - Research Site, Brick, New Jersey
  - Research Site, Florham Park, New Jersey
  - Research Site, Mineola, New York
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, San Antonio, Texas
  - Research Site, Fort Belvoir, Virginia
- Australia (7):
  - Research Site, Bedford Park
  - Research Site, Camperdown
  - Research Site, Darlinghurst
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Kurralta Park
  - Research Site, Woolloongabba
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Kortrijk
- Brazil (11):
  - Research Site, Barretos
  - Research Site, Cachoeira de Itapemirim
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Lajeado
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Research Site, Toronto, Ontario, Canada
- China (17):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Kunming
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- France (5):
  - Research Site, Bron
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Paris
- Germany (14):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Coswig
  - Research Site, Gauting
  - Research Site, Gerlingen
  - Research Site, Großhansdorf
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Homburg
  - Research Site, Immenhausen
  - Research Site, Kassel
  - Research Site, Lübeck
  - Research Site, Würzburg
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, King's Park
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- Israel (7):
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (13):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Cremona
  - Research Site, Florence
  - Research Site, Lucca
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Novara
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Roma
- Japan (22):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kitakyushu-shi
  - Research Site, Kobe
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sakaishi
  - Research Site, Sasebo-shi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Ube-shi
  - Research Site, Yokohama
  - Research Site, Yonago-shi
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Hoofddorp
  - Research Site, Zwolle
- Poland (7):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Otwock
  - Research Site, Poznan
  - Research Site, Racibórz
  - Research Site, Warsaw
  - Research Site, Wieliszew
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Focşani
  - Research Site, Iași
  - Research Site, Timișoara
- Russia (9):
  - Research Site, Arkhangelsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Pyatigorsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (10):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Elche
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Valencia
  - Research Site, Zaragoza
- Research Site, Linköping, Sweden
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Putzu City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Chiang Rai
  - Research Site, Khon Kaen
  - Research Site, Mueang
  - Research Site, Phitsanulok
  - Research Site, Songkhla
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (6):
  - Research Site, Dnipro
  - Research Site, Lviv
  - Research Site, Sumy
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Result] Herbst RS, Wu YL, Tsuboi M. Osimertinib in EGFR-Mutated Lung Cancer. Reply. N Engl J Med. 2021 Feb 18;384(7):675-676. doi: 10.1056/NEJMc2033951. No abstract available. PMID 33596365
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- [Derived] Herbst RS, John T, Grohe C, Goldman JW, Kato T, Laktionov K, Bonanno L, Tiseo M, Majem M, Domine M, Ahn MJ, Kowalski DM, Perol M, Sriuranpong V, Ozguroglu M, Bhetariya P, Markovets A, Rukazenkov Y, Muldoon C, Robichaux J, Hartmaier R, Tsuboi M, Wu YL. Molecular residual disease analysis of adjuvant osimertinib in resected EGFR-mutated stage IB-IIIA non-small-cell lung cancer. Nat Med. 2025 Jun;31(6):1958-1968. doi: 10.1038/s41591-025-03577-y. Epub 2025 Mar 17. PMID 40097663
- [Derived] Wu D, Li GF. Improving Report of the ADAURA Trial by Distinguishing Treatment-Related Adverse Events From Treatment-Emergent Adverse Events and Assessing Independence of Censoring in Final Disease-Free Survival Analyses. J Clin Oncol. 2023 Sep 10;41(26):4317-4318. doi: 10.1200/JCO.23.00604. Epub 2023 Jun 30. No abstract available. PMID 37390376
- [Derived] Tsuboi M, Herbst RS, John T, Kato T, Majem M, Grohe C, Wang J, Goldman JW, Lu S, Su WC, de Marinis F, Shepherd FA, Lee KH, Le NT, Dechaphunkul A, Kowalski D, Poole L, Bolanos A, Rukazenkov Y, Wu YL; ADAURA Investigators. Overall Survival with Osimertinib in Resected EGFR-Mutated NSCLC. N Engl J Med. 2023 Jul 13;389(2):137-147. doi: 10.1056/NEJMoa2304594. Epub 2023 Jun 4. PMID 37272535
- [Derived] John T, Grohe C, Goldman JW, Shepherd FA, de Marinis F, Kato T, Wang Q, Su WC, Choi JH, Sriuranpong V, Melotti B, Fidler MJ, Chen J, Albayaty M, Stachowiak M, Taggart S, Wu YL, Tsuboi M, Herbst RS, Majem M. Three-Year Safety, Tolerability, and Health-Related Quality of Life Outcomes of Adjuvant Osimertinib in Patients With Resected Stage IB to IIIA EGFR-Mutated NSCLC: Updated Analysis From the Phase 3 ADAURA Trial. J Thorac Oncol. 2023 Sep;18(9):1209-1221. doi: 10.1016/j.jtho.2023.05.015. Epub 2023 May 24. PMID 37236398
- [Derived] Herbst RS, Wu YL, John T, Grohe C, Majem M, Wang J, Kato T, Goldman JW, Laktionov K, Kim SW, Yu CJ, Vu HV, Lu S, Lee KY, Mukhametshina G, Akewanlop C, de Marinis F, Bonanno L, Domine M, Shepherd FA, Urban D, Huang X, Bolanos A, Stachowiak M, Tsuboi M. Adjuvant Osimertinib for Resected EGFR-Mutated Stage IB-IIIA Non-Small-Cell Lung Cancer: Updated Results From the Phase III Randomized ADAURA Trial. J Clin Oncol. 2023 Apr 1;41(10):1830-1840. doi: 10.1200/JCO.22.02186. Epub 2023 Jan 31. PMID 36720083
- [Derived] John T, Majem M, Legg D, Goldman J. Current and Future Perspectives of Health-Related Quality of Life in Resectable EGFR-Mutated Non-Small Cell Lung Cancer: A Podcast. Target Oncol. 2023 Jan;18(1):1-8. doi: 10.1007/s11523-022-00927-5. Epub 2022 Dec 19. No abstract available. PMID 36534268
- [Derived] Majem M, Goldman JW, John T, Grohe C, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Li S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Atagi S, Zeng L, Kulkarni D, Medic N, Tsuboi M, Herbst RS, Wu YL. Health-Related Quality of Life Outcomes in Patients with Resected Epidermal Growth Factor Receptor-Mutated Non-Small Cell Lung Cancer Who Received Adjuvant Osimertinib in the Phase III ADAURA Trial. Clin Cancer Res. 2022 Jun 1;28(11):2286-2296. doi: 10.1158/1078-0432.CCR-21-3530. PMID 35012927
- [Derived] Wu YL, John T, Grohe C, Majem M, Goldman JW, Kim SW, Kato T, Laktionov K, Vu HV, Wang Z, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Atasoy A, Herbst RS, Tsuboi M. Postoperative Chemotherapy Use and Outcomes From ADAURA: Osimertinib as Adjuvant Therapy for Resected EGFR-Mutated NSCLC. J Thorac Oncol. 2022 Mar;17(3):423-433. doi: 10.1016/j.jtho.2021.10.014. Epub 2021 Nov 2. PMID 34740861
- [Derived] Wu YL, Tsuboi M, John T, Grohe C, Majem M, Goldman JW, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Hodge R, Atasoy A, Rukazenkov Y, Herbst RS. A plain language summary of results from the ADAURA study: osimertinib after surgery for patients who have early-stage EGFR-mutated non-small cell lung cancer. Future Oncol. 2021 Dec 1;17(35):4827-4835. doi: 10.2217/fon-2021-0752. Epub 2021 Nov 1. PMID 34723634
- [Derived] Wu YL, Tsuboi M, He J, John T, Grohe C, Majem M, Goldman JW, Laktionov K, Kim SW, Kato T, Vu HV, Lu S, Lee KY, Akewanlop C, Yu CJ, de Marinis F, Bonanno L, Domine M, Shepherd FA, Zeng L, Hodge R, Atasoy A, Rukazenkov Y, Herbst RS; ADAURA Investigators. Osimertinib in Resected EGFR-Mutated Non-Small-Cell Lung Cancer. N Engl J Med. 2020 Oct 29;383(18):1711-1723. doi: 10.1056/NEJMoa2027071. Epub 2020 Sep 19. PMID 32955177
- [Derived] Wu YL, Herbst RS, Mann H, Rukazenkov Y, Marotti M, Tsuboi M. ADAURA: Phase III, Double-blind, Randomized Study of Osimertinib Versus Placebo in EGFR Mutation-positive Early-stage NSCLC After Complete Surgical Resection. Clin Lung Cancer. 2018 Jul;19(4):e533-e536. doi: 10.1016/j.cllc.2018.04.004. Epub 2018 May 1. PMID 29789220
- See also: Cancer — http://www.nlm.nih.gov/medlineplus/cancer.html
- See also: Lung Cancer — http://www.nlm.nih.gov/medlineplus/lungcancer.html
- See also: EGFR mutation — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&query=EGFR+mutation&x=20&y=19
- See also: Stage IB non-small cell lung cancer — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=stage+IB+non-small+cell+lung+cancer
- See also: Stage II non-small cell lung cancer — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=Stage+II+non-small+cell+lung+cancer
- See also: Stage IIIA non-small cell lung cancer — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=Stage+IIIA+non-small+cell+lung+cancer
- See also: Adjuvant chemotherapy in non-small cancer — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=adjuvant+chemotherapy+in+non-small+cancer
- See also: Complete tumour resection in non-small cancer — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=complete+tumour+resection+in+non-small+cancer
- See also: EGFR sensitivity — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=EGFR+sensitivity
- See also: EGFR inhibitors — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&v%3Asources=medlineplus-bundle&query=EGFR+inhibitors
- See also: FDA Drug and Device Resources — http://clinicaltrials.gov/ct2/info/fdalinks
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5164C00001&attachmentIdentifier=bb565084-81da-44b1-b70c-083b742cd562&fileName=SAP_redacted_D5164C00001.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5164C00001&attachmentIdentifier=e85e833e-fe2c-45c1-a278-7c9b023fd78e&fileName=D5164C00001_CSR-Synopsis.pdf&versionIdentifier=
- See also: CSR Synopsis add 1 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5164C00001&attachmentIdentifier=fe73ecf5-8e7e-4f5e-9118-e6a825cdffda&fileName=D5164C00001-CSR-addendum1-Synopsis.pdf&versionIdentifier=
- See also: CSR Synopsis add 2 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5164C00001&attachmentIdentifier=b88104d0-90ec-4a97-a0fe-f01222d612af&fileName=D5164C00001-CSR-addendum-2-Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 682 Patients were randomized to treatment at 245 Centers in 25 Countries.
Pre-assignment Details: During the 28 day screening period, participants were enrolled based on the presence of at least 1 of the 2 most frequent Epidermal growth factor receptor (EGFR) mutations in their tumor. At the time of enrolment, all participant were required to have central confirmation of EGFR mutation status per eligibility criteria (Exon 19 deletion or L858R mutation).
Groups:
- AZD9291; Placebo: Taken once daily
Period: Overall Study
Arm/Group | AZD9291 | Placebo
Started | 339 | 343
Received Treatment | 337 | 343
Completed ((Study)) | 261 | 234
Not Completed | 78 | 109
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 24 | 21
Not completed — Death | 42 | 82
Not completed — Ongoing study at data cut-off | 3 | 2
Not completed — Without specified reason | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9291 | Placebo | Total
Number analyzed (Participants) | 339 | 343 | 682
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (10.3) | 61.6 (10.5) | 62.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 248 | 478
  Male | 109 | 95 | 204
Race/Ethnicity, Customized [Number; unit: Participants]
  ASIAN (OTHER THAN CHINESE AND JAPANESE) | 77 | 65 | 142
  CHINESE | 95 | 100 | 195
  HISPANIC OR LATINO | 12 | 9 | 21
  JAPANESE | 47 | 53 | 100
  OTHER | 108 | 116 | 224
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0
  ASIAN | 216 | 218 | 434
  BLACK OR AFRICAN AMERICAN | 0 | 0 | 0
  UNKNOWN OR NOT REPORTED | 0 | 1 | 1
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0
  OTHER | 1 | 2 | 3
  WHITE | 122 | 122 | 244
Region of Enrollment [Number; unit: Participants]
  Australia | 7 | 9 | 16
  Belgium | 0 | 1 | 1
  Brazil | 8 | 6 | 14
  Canada | 1 | 3 | 4
  China | 77 | 82 | 159
  Germany | 7 | 5 | 12
  Spain | 14 | 16 | 30
  France | 4 | 5 | 9
  Hong Kong, S.A.R., China | 4 | 4 | 8
  Hungary | 1 | 1 | 2
  Israel | 9 | 3 | 12
  Italy | 15 | 17 | 32
  Japan | 46 | 53 | 99
  Poland | 4 | 9 | 13
  Romania | 2 | 2 | 4
  Russia | 43 | 39 | 82
  Sweden | 1 | 1 | 2
  Thailand | 16 | 17 | 33
  Turkey | 3 | 8 | 11
  Taiwan, China | 24 | 22 | 46
  Ukraine | 2 | 1 | 3
  United States | 13 | 8 | 21
  Viet Nam | 11 | 13 | 24
  Korea, Republic Of | 27 | 18 | 45

OUTCOME MEASURES:

1. Primary Outcome: Assess the Efficacy of AZD9291 Compared to Placebo as Measured by Disease Free Survival (DFS).
Description: Defined as the time from the date of randomization until the date of disease recurrence or death (by any cause in the absence of recurrence).
Time Frame: Up to approximately 5 years after the first patient is randomized (maximum follow up of 70 months)
Population: Full Analysis Set (FAS) stage IIA-IIIA patients
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- AZD9291 80mg Tablet; Placebo Tablet: Taken once daily
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 233 | 237
Months | 65.8 [54.4 to NA] — Insufficient DFS events to estimate upper 95% confidence interval (Kaplan Meier analysis) | 21.9 [16.6 to 27.5]
Statistical Analysis 1: Comparison: AZD9291 80mg Tablet vs Placebo Tablet; Test type: Superiority; p < 0.0001, Log Rank; Determined using a log rank test stratified by stage, race and mutation type; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.18 to 0.30] — A hazard ratio <1 favours AZD9291

2. Primary Outcome: Assess the Efficacy of AZD9291 Compared to Placebo as Measured by Disease Free Survival (DFS).
Description: as for outcome 1
Time Frame: Up to approximately 5 years after the first patient is randomized (maximum follow up of 70 months)
Population: Full Analysis Set (FAS) stage IB-IIIA patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 339 | 343
Months | 65.8 [61.7 to NA] — Insufficient DFS events to estimate upper 95% confidence interval (Kaplan Meier analysis) | 28.1 [22.1 to 35.0]
Statistical Analysis 1: Comparison: AZD9291 80mg Tablet vs Placebo Tablet; Test type: Superiority; p < 0.0001, Log Rank; Determined using a log rank test stratified by stage, race and mutation type; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.21 to 0.34] — A hazard ratio <1 favours AZD9291

3. Secondary Outcome: Disease Free Survival (DFS) Rate at 2, 3 and 5 Years
Description: Defined as the percentage of patients alive and disease free at 2, 3 and 5 years, respectively, estimated from Kaplan Meier plots of the primary endpoint of DFS.
Time Frame: Up to approximately 5 years after the first patient is randomized (maximum follow up of 70 months). DFS rate at 2 years (%), 3 years (%) and 5 years (%) are presented.
Population: Full analysis set (FAS) stage IIA-IIIA patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 233 | 237
Percentage of participants
  DFS rate at 2 years (%) | 90.0 [85.2 to 93.3] | 46.1 [39.6 to 52.4]
  DFS rate at 3 years (%) | 83.5 [77.8 to 87.8] | 33.8 [27.8 to 40.0]
  DFS rate at 5 years (%) | 53.0 [43.0 to 62.1] | 24.9 [19.0 to 31.2]

4. Secondary Outcome: Disease Free Survival (DFS) Rate at 2, 3 and 5 Years
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Full analysis set (FAS) stage IB-IIIA patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 339 | 343
Percentage of participants
  DFS rate at 2 years (%) | 90.1 [86.2 to 92.9] | 54.5 [49.0 to 59.7]
  DFS rate at 3 years (%) | 84.5 [79.9 to 88.1] | 44.4 [39.0 to 49.7]
  DFS rate at 5 years (%) | 60.9 [53.1 to 67.8] | 33.6 [28.0 to 39.2]

5. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from the date of randomization until date of death due to any cause.
Time Frame: Up to approximately 7 years after the first patient is randomized (maximum follow up of 86 months)
Population: Full Analysis Set (FAS) stage IIA-IIIA patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 233 | 237
Months | NA [NA to NA] — Insufficient OS events to estimate median and 95% confidence interval (Kaplan Meier analysis) | NA [NA to NA] — Insufficient OS events to estimate median and 95% confidence interval (Kaplan Meier analysis)
Statistical Analysis 1: Comparison: AZD9291 80mg Tablet vs Placebo Tablet; Test type: Superiority; p = 0.0004, Log Rank; Determined using a log rank test stratified by stage, race and mutation type; Hazard Ratio (HR) = 0.4913, 95.03% CI 2-sided [0.3307 to 0.7299] — A hazard ratio <1 favours AZD9291

6. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from the date of randomization until date of death due to any cause.
Time Frame: Up to approximately 7 years after the first patient is randomized (maximum follow up of 86 months)
Population: Full Analysis Set (FAS) stage IB-IIIA patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 339 | 343
Months | NA [NA to NA] — Insufficient OS events to estimate median and 95% confidence interval (Kaplan Meier analysis) | NA [NA to NA] — Insufficient OS events to estimate median and 95% confidence interval (Kaplan Meier analysis)
Statistical Analysis 1: Comparison: AZD9291 80mg Tablet vs Placebo Tablet; Test type: Superiority; p < 0.0001, Log Rank; Determined using a log rank test stratified by stage, race and mutation type; Hazard Ratio (HR) = 0.4912, 95.03% CI 2-sided [0.3439 to 0.7017] — A hazard ratio <1 favours AZD9291

7. Secondary Outcome: Overall Survival Rate at 2, 3 and 5 Years
Description: Defined as the percentage of patients alive at 2, 3 and 5 years, respectively, estimated from a Kaplan Meier plot of OS.
Time Frame: Up to approximately 7 years after the first patient is randomized (maximum follow up of 86 months). OS rate at 2 years (%), 3 years (%) and 5 years (%) are presented.
Population: Full Analysis Set (FAS) stage IIA-IIIA patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 233 | 237
Percentage of participants
  OS rate at 2 years (%) | 99.5 [96.8 to 99.9] | 92.6 [88.3 to 95.3]
  OS rate at 3 years (%) | 94.1 [90.1 to 96.5] | 85.9 [80.6 to 89.8]
  OS rate at 5 years (%) | 85.0 [79.3 to 89.2] | 72.6 [66.0 to 78.1]

8. Secondary Outcome: Overall Survival Rate at 2, 3 and 5 Years
Description: Defined as the percentage of patients alive at 2, 3 and 5 years, respectively, estimated from a Kaplan Meier plot of OS.
Time Frame: as for outcome 7
Population: Full Analysis Set (FAS) stage IB-IIIA patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 339 | 343
Percentage of participants
  OS rate at 2 years (%) | 99.4 [97.5 to 99.8] | 94.3 [91.2 to 96.3]
  OS rate at 3 years (%) | 95.3 [92.3 to 97.1] | 88.8 [84.9 to 91.8]
  OS rate at 5 years (%) | 87.6 [83.3 to 90.9] | 77.7 [72.7 to 81.9]

9. Secondary Outcome: Patient Health-related Quality of Life and Symptoms (HRQoL) by SF-36v2 Health Survey.
Description: Change from baseline will be calculated for each domain and summary scale at each scheduled post-baseline assessment. The SF-36 includes eight domains: Physical Functioning (PF); Role Limitations-Physical (RP), Vitality (VT), General Health Perceptions (GH), Bodily Pain (BP), Social Function (SF), Role Limitations-Emotional (RE), and Mental Health (MH) and two summary scores: The Physical Component Summary (PCS) and Mental Component Summary (MCS). Final scores for each scale range from 0-100 with higher scores indicating better health.
Time Frame: Measured by SF-36 Questionnaire at baseline, 12 week, 24 week and then every 24 weeks until study complete, disease recurrence or other discontinuation criteria met, up to 3 years.
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | AZD9291 80mg Tablet | Placebo Tablet
Number analyzed (Participants) | 339 | 343
Unit on a scale
  Week 12 - Bodily Pain: number analyzed (Participants) | 292 | 300
  Week 12 - Bodily Pain | 1.026 (9.448) | 1.442 (8.854)
  Week 24 - Bodily Pain: number analyzed (Participants) | 274 | 276
  Week 24 - Bodily Pain | 1.521 (9.171) | 1.462 (9.279)
  Week 48 - Bodily Pain: number analyzed (Participants) | 261 | 219
  Week 48 - Bodily Pain | 2.032 (10.226) | 2.438 (10.077)
  Week 72 - Bodily Pain: number analyzed (Participants) | 236 | 190
  Week 72 - Bodily Pain | 2.471 (9.787) | 2.335 (9.566)
  Week 96 - Bodily Pain: number analyzed (Participants) | 227 | 165
  Week 96 - Bodily Pain | 2.326 (10.865) | 2.921 (10.153)
  Week 120 - Bodily Pain: number analyzed (Participants) | 218 | 152
  Week 120 - Bodily Pain | 2.906 (10.181) | 2.778 (11.295)
  Week 144 - Bodily Pain: number analyzed (Participants) | 200 | 132
  Week 144 - Bodily Pain | 3.045 (11.410) | 3.324 (10.258)
  Week 156 - Bodily Pain: number analyzed (Participants) | 179 | 106
  Week 156 - Bodily Pain | 2.552 (11.994) | 3.116 (10.692)
  Week 12 - General Health Perceptions: number analyzed (Participants) | 294 | 303
  Week 12 - General Health Perceptions | -0.597 (8.319) | 0.343 (7.497)
  Week 24 - General Health Perceptions: number analyzed (Participants) | 279 | 277
  Week 24 - General Health Perceptions | -0.079 (8.910) | 0.763 (8.122)
  Week 48 - General Health Perceptions: number analyzed (Participants) | 264 | 220
  Week 48 - General Health Perceptions | 0.103 (8.029) | 1.042 (8.416)
  Week 72 - General Health Perceptions: number analyzed (Participants) | 239 | 191
  Week 72 - General Health Perceptions | 0.275 (7.958) | 2.339 (8.197)
  Week 96 - General Health Perceptions: number analyzed (Participants) | 230 | 165
  Week 96 - General Health Perceptions | -0.119 (8.195) | 1.818 (7.903)
  Week 120 - General Health Perceptions: number analyzed (Participants) | 221 | 152
  Week 120 - General Health Perceptions | -0.368 (8.461) | 0.964 (8.518)
  Week 144 - General Health Perceptions: number analyzed (Participants) | 202 | 132
  Week 144 - General Health Perceptions | 0.209 (8.671) | 1.342 (8.789)
  Week 156 - General Health Perceptions: number analyzed (Participants) | 183 | 106
  Week 156 - General Health Perceptions | -0.128 (8.987) | 2.166 (8.670)
  Week 12 - Mental Health: number analyzed (Participants) | 291 | 302
  Week 12 - Mental Health | 0.928 (8.538) | 1.892 (8.497)
  Week 24 - Mental Health: number analyzed (Participants) | 276 | 277
  Week 24 - Mental Health | 1.249 (8.780) | 1.275 (9.660)
  Week 48 - Mental Health: number analyzed (Participants) | 262 | 219
  Week 48 - Mental Health | 2.456 (8.920) | 2.234 (8.676)
  Week 72 - Mental Health: number analyzed (Participants) | 237 | 190
  Week 72 - Mental Health | 1.540 (9.029) | 2.011 (8.954)
  Week 96 - Mental Health: number analyzed (Participants) | 228 | 165
  Week 96 - Mental Health | 1.352 (8.560) | 2.101 (8.986)
  Week 120 - Mental Health: number analyzed (Participants) | 219 | 152
  Week 120 - Mental Health | 0.723 (9.738) | 2.307 (10.139)
  Week 144 - Mental Health: number analyzed (Participants) | 200 | 132
  Week 144 - Mental Health | 0.517 (9.609) | 1.428 (8.914)
  Week 156 - Mental Health: number analyzed (Participants) | 180 | 106
  Week 156 - Mental Health | 0.386 (10.215) | 2.000 (9.651)
  Week 12 - Physical functioning: number analyzed (Participants) | 294 | 302
  Week 12 - Physical functioning | -0.314 (6.762) | 0.898 (6.646)
  Week 24 - Physical functioning: number analyzed (Participants) | 277 | 275
  Week 24 - Physical functioning | 0.494 (6.783) | 0.923 (7.014)
  Week 48 - Physical functioning: number analyzed (Participants) | 263 | 220
  Week 48 - Physical functioning | 0.940 (7.595) | 1.914 (7.899)
  Week 72 - Physical functioning: number analyzed (Participants) | 238 | 191
  Week 72 - Physical functioning | 1.079 (6.725) | 2.042 (7.283)
  Week 96 - Physical functioning: number analyzed (Participants) | 229 | 165
  Week 96 - Physical functioning | 0.637 (8.220) | 2.016 (7.048)
  Week 120 - Physical functioning: number analyzed (Participants) | 220 | 152
  Week 120 - Physical functioning | 1.449 (7.207) | 2.540 (7.424)
  Week 144 - Physical functioning: number analyzed (Participants) | 202 | 132
  Week 144 - Physical functioning | 1.869 (6.767) | 1.939 (8.238)
  Week 156 - Physical functioning: number analyzed (Participants) | 182 | 105
  Week 156 - Physical functioning | 0.997 (7.537) | 2.187 (8.293)
  Week 12 - Role Limitations - Emotional: number analyzed (Participants) | 292 | 303
  Week 12 - Role Limitations - Emotional | 0.381 (10.413) | 2.333 (11.168)
  Week 24 - Role Limitations - Emotional: number analyzed (Participants) | 276 | 276
  Week 24 - Role Limitations - Emotional | 0.858 (11.317) | 1.678 (11.571)
  Week 48 - Role Limitations - Emotional: number analyzed (Participants) | 262 | 220
  Week 48 - Role Limitations - Emotional | 2.179 (11.131) | 2.628 (10.952)
  Week 72 - Role Limitations - Emotional: number analyzed (Participants) | 237 | 191
  Week 72 - Role Limitations - Emotional | 1.410 (11.861) | 1.860 (11.424)
  Week 96 - Role Limitations - Emotional: number analyzed (Participants) | 227 | 165
  Week 96 - Role Limitations - Emotional | 1.657 (12.405) | 1.899 (12.379)
  Week 120 - Role Limitations - Emotional: number analyzed (Participants) | 219 | 152
  Week 120 - Role Limitations - Emotional | 1.765 (11.966) | 2.360 (12.663)
  Week 144 - Role Limitations - Emotional: number analyzed (Participants) | 200 | 132
  Week 144 - Role Limitations - Emotional | 1.654 (12.081) | 2.532 (13.113)
  Week 156 - Role Limitations - Emotional: number analyzed (Participants) | 181 | 106
  Week 156 - Role Limitations - Emotional | 0.519 (12.351) | 2.201 (13.022)
  Week 12 - Role Limitations - Physical: number analyzed (Participants) | 292 | 303
  Week 12 - Role Limitations - Physical | 1.056 (9.263) | 2.915 (8.977)
  Week 24 - Role Limitations - Physical: number analyzed (Participants) | 277 | 276
  Week 24 - Role Limitations - Physical | 1.727 (10.265) | 4.063 (9.295)
  Week 48 - Role Limitations - Physical: number analyzed (Participants) | 262 | 220
  Week 48 - Role Limitations - Physical | 3.437 (10.592) | 5.332 (9.663)
  Week 72 - Role Limitations - Physical: number analyzed (Participants) | 237 | 191
  Week 72 - Role Limitations - Physical | 3.581 (11.037) | 5.424 (9.670)
  Week 96 - Role Limitations - Physical: number analyzed (Participants) | 228 | 165
  Week 96 - Role Limitations - Physical | 3.240 (10.807) | 5.321 (9.997)
  Week 120 - Role Limitations - Physical: number analyzed (Participants) | 219 | 152
  Week 120 - Role Limitations - Physical | 4.717 (11.238) | 5.348 (11.395)
  Week 144 - Role Limitations - Physical: number analyzed (Participants) | 200 | 132
  Week 144 - Role Limitations - Physical | 3.525 (10.860) | 5.444 (10.547)
  Week 156 - Role Limitations - Physical: number analyzed (Participants) | 181 | 106
  Week 156 - Role Limitations - Physical | 3.151 (11.378) | 5.572 (10.954)
  Week 12 - Social Function: number analyzed (Participants) | 292 | 301
  Week 12 - Social Function | 1.391 (9.615) | 3.164 (9.171)
  Week 24 - Social Function: number analyzed (Participants) | 276 | 276
  Week 24 - Social Function | 2.634 (9.526) | 3.433 (10.348)
  Week 48 - Social Function: number analyzed (Participants) | 262 | 220
  Week 48 - Social Function | 3.731 (9.919) | 4.170 (10.156)
  Week 72 - Social Function: number analyzed (Participants) | 237 | 190
  Week 72 - Social Function | 3.025 (10.094) | 4.802 (10.351)
  Week 96 - Social Function: number analyzed (Participants) | 228 | 165
  Week 96 - Social Function | 3.651 (10.011) | 4.405 (10.790)
  Week 120 - Social Function: number analyzed (Participants) | 219 | 152
  Week 120 - Social Function | 3.297 (10.723) | 4.386 (11.355)
  Week 144 - Social Function: number analyzed (Participants) | 200 | 132
  Week 144 - Social Function | 2.582 (10.638) | 3.912 (10.929)
  Week 156 - Social Function: number analyzed (Participants) | 180 | 106
  Week 156 - Social Function | 2.423 (10.658) | 4.351 (12.144)
  Week 12 - Vitality: number analyzed (Participants) | 290 | 302
  Week 12 - Vitality | 0.570 (7.987) | 2.344 (8.207)
  Week 24 - Vitality: number analyzed (Participants) | 275 | 277
  Week 24 - Vitality | 0.630 (8.996) | 2.463 (9.461)
  Week 48 - Vitality: number analyzed (Participants) | 261 | 219
  Week 48 - Vitality | 2.231 (9.209) | 3.029 (8.972)
  Week 72 - Vitality: number analyzed (Participants) | 236 | 190
  Week 72 - Vitality | 1.082 (9.387) | 3.815 (8.869)
  Week 96 - Vitality: number analyzed (Participants) | 228 | 165
  Week 96 - Vitality | 1.147 (9.052) | 3.474 (9.071)
  Week 120 - Vitality: number analyzed (Participants) | 219 | 152
  Week 120 - Vitality | 1.139 (9.458) | 3.224 (9.122)
  Week 144 - Vitality: number analyzed (Participants) | 200 | 132
  Week 144 - Vitality | 0.386 (9.724) | 2.070 (9.285)
  Week 156 - Vitality: number analyzed (Participants) | 180 | 106
  Week 156 - Vitality | 0.825 (9.342) | 2.970 (8.831)
  Week 12 - Mental Component Summary: number analyzed (Participants) | 291 | 301
  Week 12 - Mental Component Summary | 0.986 (8.068) | 2.603 (8.965)
  Week 24 - Mental Component Summary: number analyzed (Participants) | 274 | 275
  Week 24 - Mental Component Summary | 1.333 (8.919) | 1.936 (10.152)
  Week 48 - Mental Component Summary: number analyzed (Participants) | 261 | 219
  Week 48 - Mental Component Summary | 2.788 (9.301) | 2.757 (9.141)
  Week 72 - Mental Component Summary: number analyzed (Participants) | 236 | 190
  Week 72 - Mental Component Summary | 1.434 (9.635) | 2.577 (9.116)
  Week 96 - Mental Component Summary: number analyzed (Participants) | 227 | 165
  Week 96 - Mental Component Summary | 1.823 (9.439) | 2.415 (10.023)
  Week 120 - Mental Component Summary: number analyzed (Participants) | 218 | 152
  Week 120 - Mental Component Summary | 1.027 (10.286) | 2.554 (10.548)
  Week 144 - Mental Component Summary: number analyzed (Participants) | 200 | 132
  Week 144 - Mental Component Summary | 0.580 (9.994) | 1.870 (9.857)
  Week 156 - Mental Component Summary: number analyzed (Participants) | 179 | 106
  Week 156 - Mental Component Summary | 0.322 (10.077) | 2.269 (10.647)
  Week 12 - Physical Component Summary: number analyzed (Participants) | 291 | 301
  Week 12 - Physical Component Summary | 0.161 (6.341) | 1.144 (6.078)
  Week 24 - Physical Component Summary: number analyzed (Participants) | 274 | 275
  Week 24 - Physical Component Summary | 0.878 (7.009) | 1.938 (6.643)
  Week 48 - Physical Component Summary: number analyzed (Participants) | 261 | 219
  Week 48 - Physical Component Summary | 1.356 (6.800) | 2.797 (7.497)
  Week 72 - Physical Component Summary: number analyzed (Participants) | 236 | 190
  Week 72 - Physical Component Summary | 1.989 (6.941) | 3.360 (6.985)
  Week 96 - Physical Component Summary: number analyzed (Participants) | 227 | 165
  Week 96 - Physical Component Summary | 1.497 (7.591) | 3.343 (6.792)
  Week 120 - Physical Component Summary: number analyzed (Participants) | 218 | 152
  Week 120 - Physical Component Summary | 2.611 (7.291) | 3.175 (8.210)
  Week 144 - Physical Component Summary: number analyzed (Participants) | 200 | 132
  Week 144 - Physical Component Summary | 2.635 (7.374) | 3.353 (8.042)
  Week 156 - Physical Component Summary: number analyzed (Participants) | 179 | 105
  Week 156 - Physical Component Summary | 2.133 (7.909) | 3.644 (8.731)

10. Secondary Outcome: Plasma Concentrations of AZD9291
Description: The pharmacokinetics exposure parameters derived from plasma concentrations of AZD9291
Time Frame: Collected at pre-dose, 0.5-1.5hours and 2-4hours post-dose up to 96 weeks (approximately 24 months)
Population: Pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | AZD9291 80mg Tablet
Number analyzed (Participants) | 325
nM
  Week 4 - Pre-dose: number analyzed (Participants) | 247
  Week 4 - Pre-dose | 380.2563 (60.4465)
  Week 4 - 0.5-1.5 hours: number analyzed (Participants) | 246
  Week 4 - 0.5-1.5 hours | 383.9142 (74.3191)
  Week 4 - 2-4 hours: number analyzed (Participants) | 246
  Week 4 - 2-4 hours | 463.0098 (56.3562)
  Week 24- Pre-dose: number analyzed (Participants) | 213
  Week 24- Pre-dose | 288.8266 (181.8255)
  Week 24 - 0.5-1.5 hours: number analyzed (Participants) | 212
  Week 24 - 0.5-1.5 hours | 303.8269 (116.9411)
  Week 24 - 2-4 hours: number analyzed (Participants) | 211
  Week 24 - 2-4 hours | 358.831 (116.0567)
  Week 48- Pre-dose: number analyzed (Participants) | 198
  Week 48- Pre-dose | 301.7346 (125.4901)
  Week 48 - 0.5-1.5 hours: number analyzed (Participants) | 196
  Week 48 - 0.5-1.5 hours | 311.3503 (101.1574)
  Week 48 - 2-4 hours: number analyzed (Participants) | 195
  Week 48 - 2-4 hours | 375.6666 (69.9838)
  Week 96- Pre-dose: number analyzed (Participants) | 126
  Week 96- Pre-dose | 287.5375 (95.6634)
  Week 96 - 0.5-1.5 hours: number analyzed (Participants) | 127
  Week 96 - 0.5-1.5 hours | 273.3198 (126.003)
  Week 96 - 2-4 hours: number analyzed (Participants) | 127
  Week 96 - 2-4 hours | 341.5805 (79.0578)

11. Secondary Outcome: Plasma Concentrations of AZ5104 Metabolites
Description: The pharmacokinetics exposure parameters derived from plasma concentrations of AZ5104 metabolites
Time Frame: From date of dosing to week 96 (approximately 24 months)
Population: Pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- AZ5104: AZD9291 metabolite
Arm/Group | AZ5104
Number analyzed (Participants) | 325
nM
  Week 4 - Pre-dose: number analyzed (Participants) | 247
  Week 4 - Pre-dose | 44.4619 (66.2108)
  Week 4 - 0.5-1.5 hours: number analyzed (Participants) | 246
  Week 4 - 0.5-1.5 hours | 45.2280 (67.0500)
  Week 4 - 2-4 hours: number analyzed (Participants) | 246
  Week 4 - 2-4 hours | 49.6081 (65.5757)
  Week 24 - Pre-dose: number analyzed (Participants) | 213
  Week 24 - Pre-dose | 38.7314 (111.0996)
  Week 24 - 0.5-1.5 hours: number analyzed (Participants) | 212
  Week 24 - 0.5-1.5 hours | 39.1687 (86.1118)
  Week 24 - 2-4 hours: number analyzed (Participants) | 211
  Week 24 - 2-4 hours | 41.3251 (99.2633)
  Week 48 - Pre-dose: number analyzed (Participants) | 198
  Week 48 - Pre-dose | 41.1778 (53.8923)
  Week 48 - 0.5-1.5 hours: number analyzed (Participants) | 196
  Week 48 - 0.5-1.5 hours | 40.9276 (53.9916)
  Week 48 - 2-4 hours: number analyzed (Participants) | 195
  Week 48 - 2-4 hours | 42.9143 (68.8102)
  Week 96 - Pre-dose: number analyzed (Participants) | 126
  Week 96 - Pre-dose | 38.0205 (81.4442)
  Week 96 - 0.5-1.5 hours: number analyzed (Participants) | 127
  Week 96 - 0.5-1.5 hours | 36.9723 (101.2317)
  Week 96 - 2-4 hours: number analyzed (Participants) | 127
  Week 96 - 2-4 hours | 39.8057 (78.0300)

12. Secondary Outcome: Plasma Concentrations of AZ7550 Metabolites
Description: The pharmacokinetics exposure parameters derived from plasma concentrations of AZ7550 metabolites
Time Frame: From date of dosing to week 96 (approximately 24 months)
Population: Pharmacokinetic analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- AZ7550: AZD9291 metabolite
Arm/Group | AZ7550
Number analyzed (Participants) | 325
nM
  Week 4 - Pre-dose: number analyzed (Participants) | 225
  Week 4 - Pre-dose | 44.3492 (56.5153)
  Week 4 - 0.5-1.5 hours: number analyzed (Participants) | 224
  Week 4 - 0.5-1.5 hours | 44.7386 (55.0410)
  Week 4 - 2-4 hours: number analyzed (Participants) | 223
  Week 4 - 2-4 hours | 48.0864 (61.8700)
  Week 24 - Pre-dose: number analyzed (Participants) | 171
  Week 24 - Pre-dose | 40.7113 (75.3663)
  Week 24 - 0.5-1.5 hours: number analyzed (Participants) | 170
  Week 24 - 0.5-1.5 hours | 40.9375 (65.8656)
  Week 24 - 2-4 hours: number analyzed (Participants) | 169
  Week 24 - 2-4 hours | 44.1476 (60.2684)
  Week 48 - Pre-dose: number analyzed (Participants) | 104
  Week 48 - Pre-dose | 41.3862 (52.2259)
  Week 48 - 0.5-1.5 hours: number analyzed (Participants) | 103
  Week 48 - 0.5-1.5 hours | 41.0467 (52.9773)
  Week 48 - 2-4 hours: number analyzed (Participants) | 102
  Week 48 - 2-4 hours | 40.4486 (99.6574)
  Week 96 - Pre-dose: number analyzed (Participants) | 30
  Week 96 - Pre-dose | 28.1890 (180.0937)
  Week 96 - 0.5-1.5 hours: number analyzed (Participants) | 31
  Week 96 - 0.5-1.5 hours | 30.2419 (155.4156)
  Week 96 - 2-4 hours: number analyzed (Participants) | 31
  Week 96 - 2-4 hours | 33.9653 (79.2841)

ADVERSE EVENTS:
Time Frame: Adverse events with onset date on or after the date of first dose up to and including 28 days following discontinuation of study treatment and before starting subsequent cancer therapy, up to approximately 3 years. All-Cause Mortality assessed up to approximately 7 years.
Description: Please note the "All-Cause Mortality" section has more subjects at risk because it is based off of the Full Analysis Set, which includes all randomized participants.
  The remainder of the AE sections are based off the Safety Analysis Set, which includes all patients who received at least 1 dose of study treatment.
Groups:
- AZD9291; Placebo: Description (Arm-group)
Arm/Group | AZD9291 | Placebo
All-Cause Mortality (participants affected / at risk) | 42/339 | 82/343
Serious Adverse Events (participants affected / at risk) | 68/337 | 47/343
Other Adverse Events (participants affected / at risk) | 312/337 | 262/343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 (N=337) | Placebo (N=343)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (6) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Otolithiasis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 (N=337) | Placebo (N=343)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 (29) | 5 (5)
Dizziness (Nervous system disorders) | 28 (38) | 27 (31)
Headache (Nervous system disorders) | 27 (31) | 33 (49)
Insomnia (Psychiatric disorders) | 18 (20) | 17 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 66 (86) | 61 (74)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (22) | 8 (8)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 41 (49) | 16 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 84 (95) | 23 (25)
Nail disorder (Skin and subcutaneous tissue disorders) | 22 (22) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 70 (88) | 30 (42)
Rash (Skin and subcutaneous tissue disorders) | 34 (47) | 12 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22 (29) | 14 (20)
Skin fissures (Skin and subcutaneous tissue disorders) | 19 (26) | 0 (0)
Hypertension (Vascular disorders) | 14 (16) | 18 (21)
Dry eye (Eye disorders) | 20 (20) | 12 (20)
Anaemia (Blood and lymphatic system disorders) | 28 (41) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 20 (25) | 5 (6)
Constipation (Gastrointestinal disorders) | 21 (29) | 18 (21)
Diarrhoea (Gastrointestinal disorders) | 158 (309) | 71 (114)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 18 (20) | 14 (14)
Leukopenia (Blood and lymphatic system disorders) | 20 (44) | 6 (6)
Mouth ulceration (Gastrointestinal disorders) | 39 (82) | 10 (16)
Nausea (Gastrointestinal disorders) | 34 (37) | 19 (20)
Stomatitis (Gastrointestinal disorders) | 59 (102) | 15 (17)
Toothache (Gastrointestinal disorders) | 8 (10) | 18 (25)
Vomiting (Gastrointestinal disorders) | 30 (43) | 16 (20)
Asthenia (General disorders) | 18 (21) | 17 (27)
Fatigue (General disorders) | 32 (45) | 18 (20)
Neutropenia (Blood and lymphatic system disorders) | 21 (31) | 1 (1)
Bronchitis (Infections and infestations) | 12 (16) | 18 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (47) | 0 (0)
Conjunctivitis (Infections and infestations) | 18 (25) | 10 (11)
Influenza (Infections and infestations) | 21 (28) | 15 (16)
Nasopharyngitis (Infections and infestations) | 50 (118) | 36 (74)
Paronychia (Infections and infestations) | 92 (145) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 53 (83) | 38 (54)
Urinary tract infection (Infections and infestations) | 24 (31) | 16 (21)
Alanine aminotransferase increased (Investigations) | 21 (31) | 26 (37)
Aspartate aminotransferase increased (Investigations) | 22 (32) | 27 (33)
Blood creatinine increased (Investigations) | 31 (41) | 7 (9)
Electrocardiogram qt prolonged (Investigations) | 30 (49) | 8 (9)
Neutrophil count decreased (Investigations) | 26 (48) | 3 (4)
Platelet count decreased (Investigations) | 21 (36) | 2 (3)
Weight decreased (Investigations) | 35 (40) | 9 (10)
White blood cell count decreased (Investigations) | 25 (53) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 49 (55) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (26) | 37 (42)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (28) | 26 (37)

LIMITATIONS AND CAVEATS:
Primary analysis was performed two years early as per IDMC recommendation and the exploratory analysis of final DFS data at the prespecified maturity of approx. 50% was done in 2022. After the final DFS data analysis and until the final OS analysis, only limited data were collected: subsequent anti-cancer treatment, survival status and limited safety data. The AZ7550 metabolite samples were not analyzed after Mar 2019, so the ratio of metabolite to AZD9291 was not available for calculation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT02511106/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT02511106/SAP_001.pdf